CLINICAL TRIAL: NCT02347852
Title: Assessment of Physical Activity During Therapy With Regorafenib for Metastatic Colorectal Cancer
Acronym: REGO-ACT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17816; SV1415AT (Other: Company internal)
Record Dates: First submitted 2014-12-22; First posted 2015-01-27 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Physical activity / Cohort 1: The non influenced and non triggered habitual physical activity of patients will be assessed by pedometer and physical activity questionnaire. The study population will consist of patients with metastatic CRC (mCRC) who are included in the NIS CORRELATE, have been previously treated with other approved regimens for metastatic disease and for whom a decision has been made by the physician to treat with regorafenib according to local health authority approved label prior to and independent of the inclusion into this observational study.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Stivarga is available as tablets (40 mg). It is taken in four-week treatment cycles at a recommended starting dose of 160 mg once every day for three weeks, followed by a week off.

SUMMARY:
The purpose of this trial is to quantitatively assess the average amount of physical activity that patients are capable to perform while receiving regorafenib for the treatment of metastatic colorectal cancer. The assessment of this reference value, measured by CE (Conformité Européene)-certified pedometer and international physical activity questionnaire, will allow an estimation on the feasible amount of physical activity for patients in this therapeutic setting.

This study is available for patients who are included in the global non-interventional study CORRELATE (Safety and efficacy of regorafenib in metastatic colorectal cancer patients; NCT01843400) in Austria.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mCRC who have been previously treated with, or are not considered candidates for, other locally approved standard treatment(s) and for whom the decision has been made per investigator's routine treatment practice to prescribe regorafenib.
* Patients enrolled in NIS CORRELATE in Austria
* Signed patient informed consent for local OS

Exclusion Criteria:

* Subjects unwilling to complete all questionnaires involved in the local OS
* Subjects unwilling to wear the pedometer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of NIS CORRELATE (NCT02042144, Safety and Effectiveness of Regorafenib in Routine Clinical Practice Settings) in Austria
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

PRIMARY OUTCOMES:
Amount of physical activity assessed by a pedometer (smartLAB) and an international physical activity questionnaire | At 3 months

SECONDARY OUTCOMES:
Relation of the amount of physical activity to QoL (Quality of Life) data assessed in CORRELATE (NCT02042144, 'Safety and Effectiveness of Regorafenib in Routine Clinical Practice Settings') | At 3 months
Relation of the amount of physical activity to fatigue data assessed in CORRELATE (NCT02042144, 'Safety and Effectiveness of Regorafenib in Routine Clinical Practice Settings') | At 3 months
Relation of the amount of physical activity to DCR (Disease Control Rate) data assessed in CORRELATE (NCT02042144, 'Safety and Effectiveness of Regorafenib in Routine Clinical Practice Settings') | At 3 months
Relation of the amount of physical activity to OS (Overall Survival) data assessed in CORRELATE (NCT02042144, 'Safety and Effectiveness of Regorafenib in Routine Clinical Practice Settings') | At 3 months
Relation of the amount of physical activity to PFS (Progression Free Survival) data assessed in CORRELATE (NCT02042144, 'Safety and Effectiveness of Regorafenib in Routine Clinical Practice Settings') | At 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Klinikum Kreuzschwestern Wels GmbH, Multiple Locations, Austria